CLINICAL TRIAL: NCT05774795
Title: LOng-Term Fate of Moderate Aortic Regurgitation Left Untreated at the Time of Mitral Valve Surgery
Status: Completed | Type: Observational
Sponsor: Michele De Bonis (Other)
Responsible Party: Sponsor-Investigator, Michele De Bonis, Chief of Cardiac Surgery of the Advanced and Research Therapies, Ospedale San Raffaele
Organization: Ospedale San Raffaele (Other)
Other Study IDs: LOTMAR
Record Dates: First submitted 2023-01-30; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Aortic Regurgitation; Mitral Regurgitation
MeSH Terms: conditions — Aortic Valve Insufficiency; Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mitral valve surgery only
  Interventions: Procedure: Mitral valve surgery
- Mitral valve surgery + Aortic valve surgery
  Interventions: Procedure: Mitral valve surgery; Procedure: Aortic valve surgery

INTERVENTIONS:
Procedure: Mitral valve surgery — Mitral valve repair or replacement to treat mitral regurgitation
Procedure: Aortic valve surgery — Aortic valve replacement to treat aortic regurgitation
  Groups: Mitral valve surgery + Aortic valve surgery

SUMMARY:
Multivalvular heart disease is a highly prevalent clinical condition that comprises 14.6% of the patients undergoing valvular surgery. Specifically, aortic valve regurgitation (AR) can be present in a considerable proportion of patients undergoing mitral valve (MV) surgery. In the Society of Thoracic Surgeons database, con- comitant aortic and mitral surgery accounted for 57.8% of the total multivalvular procedures with an unadjusted mortality rate of 10.7%.

When both the aortic and MVs exhibit severe disease, con- comitant valve surgery is well-accepted by the surgical commu- nity and supported by current guidelines. On the other hand, when the aortic valve (AV) shows only moderate regurgita- tion, which would not be surgically treated if singly present, the appropriate management of the AV pathology at the time of MV surgery is still under debate.

The American College of Cardiology guidelines state that aortic valve replacement (AVR) is reasonable (class IIa) in patients with moderate AR (stage B) while undergoing surgery on the ascend- ing aorta, a coronary artery bypass graft or MV surgery (level of evidence: C). Conversely, the latest European Society of Cardiology guidelines on valvular heart disease define as con- troversial the decision to treat the AV in patients with moderate AR who undergo MV surgery, considering the slow progression of this disease. In this group of patients, they advocate a heart team approach that will take into account the aetiology of AR, the life expectancy of the patient, the operative risk and other clinical factors.

This disagreement may lead to uncertainty about how patients with less than severe AR should be managed during MV surgery, especially considering the burden of double-valve surgical procedures.

The goal of this study is to evaluate the immediate and long- term outcomes, including the need for a new procedure on the AV, in patients with moderate AR at the time of MV surgery.

ELIGIBILITY:
Inclusion Criteria:

General criteria for both groups

* Adult patients;
* Patients undergoing mitral valve surgery, with moderate-grade AR, as assessed by preoperative echocardiography;

Specific criteria Group 1 (study group) - Patients who have not undergone aortic valve surgery in conjunction with mitral valve surgery

Specific criteria Group 2 (control group)

- Patients undergoing aortic valve surgery in conjunction with mitral valve surgery

Exclusion Criteria:

* Patients who have not undergone mitral surgery
* Patients undergoing multivalvular surgery other than mitro-aortic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients needing a mitral valve surgery and affected by moderate aortic regurgitation. In one group, also aortic valve surgery is performed, in the other, only surgery on the mitral valve is performed
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Mortality | through study completion, an average of 12 years

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No